CLINICAL TRIAL: NCT02860260
Title: Kinetics of Plasma and Serum Levels of Brain-Derived Neurotrophic Factor (BDNF) in Patients With Ischemic Stroke: Effect of Intravenous Fibrinolysis With Rt-PA
Brief Title: Kinetics of Plasma and Serum Levels of Brain-Derived Neurotrophic Factor (BDNF) in Patients With Ischemic Stroke
Acronym: BDNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: BEJOT
Record Dates: First submitted 2016-08-01; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: Ischemic Stroke
Keywords: BDNF
MeSH Terms: conditions — Ischemic Stroke | interventions — Blood Specimen Collection

ARMS (2):
- Patients with fibrinolysis (Experimental)
  Interventions: Biological: Blood samples; Other: Cerebral MRI
- Patients without fibrinolysis (Placebo Comparator)
  Interventions: Biological: Blood samples; Other: Cerebral MRI

INTERVENTIONS:
Biological: Blood samples
Other: Cerebral MRI

SUMMARY:
The aim of this study is to show for the first time that treatment with intravenous fibrinolysis using rt-PA in patients with recent ischemic stroke is accompanied by increases in circulating levels of BDNF, which may reflect an increase in BDNF synthesis in the brain.

The analysis of the recovery of functional and cognitive abilities as well as mood at 3 months will allow us to study the impact of BDNF on these parameters. Thus, depending on the results obtained, circulating BDNF could serve as an early marker of these.

ELIGIBILITY:
Inclusion Criteria:

* Patients (or their person of trust in cases of inability) who have been informed about the research and given their consent to take part
* Patients aged 18 years or older
* Patients who have suffered a de novo recent ischemic stroke < 12 hours
* Patients who had cerebral imaging (CT-Scan or MRI)
* Ischemic stroke severity, measured by the National Institute of Health Stroke Score (NIHSS), between 4 and 20

Exclusion Criteria:

Patients without national health insurance cover

* Patients with a clinical history of stroke
* Patients with cerebral or sub-arachnoid haemorrhage
* Patients with a transient ischemic attack
* Time of symptom onset unknown
* Patients with severe aphasia at the time of the ischemic stroke defined by a sub-score for item 9 (best language) of the NIHSS ≥ 2
* Patients with dementia prior to the ischemic stroke
* Patients with a significant loss of autonomy prior to the ischemic stroke, defined by a Rankin score ≥ 4
* Patients with aphasia before the ischemic stroke
* Patients with a contra-indication for cerebral MRI
* Pregnant or breast-feeding women
* Adults under guardianship
* Subjects in custody
* Patients who do not speak French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Measurement of plasma levels of BDNF | Change from baseline at Day1, Day 7 and Month 3
Measurement of serum levels of BDNF | Change from baseline at Day1, Day 7 and Month 3

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Dijon, France